CLINICAL TRIAL: NCT05036109
Title: DAILY: Vitamin D, Aspirin, ExercIse, Low Saturated Fat Foods StudY in Colorectal Cancer Patients With Minimal Residual Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0320; NCI-2021-09193 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Aspirin; Vitamin D; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aspirin, Vitamin D (Other): by mouth every day for up to 90 days
  Interventions: Drug: Aspirin; Drug: Vitamin D; Dietary Supplement: Diet; Other: Physical Activity; Behavioral: Behavioral Support Counseling Sessions

INTERVENTIONS:
Drug: Aspirin — by mouth every day for up to 90 days
Drug: Vitamin D — by mouth every day for up to 90 days
Dietary Supplement: Diet — Patients will receive counseling promoting a plant-based diet and avoidance of Western dietary patterns in a one on one session with a licensed dietitian prior to day 1.
Other: Physical Activity — The exercise goal is to increase recreational physical activity from baseline by at least 10 MET hours per week, which is equivalent to 150 minutes of moderate activity weekly
Behavioral: Behavioral Support Counseling Sessions — Patients will undergo a one-on-one counseling session prior to day 1

SUMMARY:
To learn if lifestyle changes (such as diet and exercise) combined with daily aspirin and vitamin D can affect the likelihood of advanced colorectal cancer coming back (recurring)

DETAILED DESCRIPTION:
Primary Objective:

To estimate the ctDNA clearance rate of colorectal cancer participants with minimal residual disease after 3 months of optimal lifestyle interventions

Secondary Objectives:

* To evaluate the dynamics of ctDNA allele fractions after 3 months of optimal lifestyle interventions and every 3 months thereafter up to 12 months
* To estimate the recurrence rate at 1 year in subjects who complete 3 months of optimal lifestyle interventions

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of study entry
* ECOG 0-1
* Histologically documented high-risk stage II, stage III, or stage IV colorectal adenocarcinoma with no evidence of disease following definitive local therapy (including surgical resection or ablation)
* No radiographic evidence of disease by contrast enhanced CT chest/abdomen/pelvis
* Presence of detectable ctDNA mutation that matches mutations found in tumor tissue
* Completion of all standard of care adjuvant therapy
* Platelet count >50,000
* Ability to give informed consent
* Ability to complete all questionnaires involved in study

Exclusion Criteria:

* Concurrent malignancy under active treatment
* Known active gastrointestinal bleeding or peptic ulcer disease
* Known hypersensitivity to vitamin D or aspirin
* CrCl<30 mL/min within 30 days of starting the intervention
* Current usage of therapeutic anticoagulation (warfarin, Eliquis, Xarelto)
* Inability to safely participate in physical activity in the opinion of the treating oncologist
* Pregnant or nursing women. N.B.: urine pregnancy test will be administered as part of the screening process.
* Persistent hypercalcemia or conditions predisposing to hypercalcemia (i.e., hyperparathyroidism)
* Known symptomatic genitourinary stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-02-04 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
To estimate the ctDNA clearance rate of colorectal cancer patients with minimal residual disease | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alisha Bent, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT05036109/ICF_000.pdf